CLINICAL TRIAL: NCT01140646
Title: Phase II Evaluation of S-Adenosyl-L-Methionine (SAMe) for the Treatment of Hot Flashes
Brief Title: Evaluation of SAMe for Hot Flashes
Acronym: SAMe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC09C4; NCI-2010-01224 (Registry Identifier: NCI's CTRO); MC09C4 (Other: Mayo Clinic Cancer Center); 10-001896 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Healthy, no Evidence of Disease; Hot Flashes
Keywords: Hot flashes, dietary supplements, symptom management
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): The first week of the study is a baseline week where data are being collected but study agent is not being taken. Patients then receive oral s-adenosyl-L-methionine, 400 mg, once daily on days 8-14 and twice daily on days 15-49 in the absence of unacceptable toxicity.
  Interventions: Drug: S-adenosyl-L-methionine disulfate p-toluene-sulfonate; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: S-adenosyl-L-methionine disulfate p-toluene-sulfonate — Given orally
  Other Names: SAMe disulfate p-toluene-sulfonate
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: S-adenosyl-L-methionine may help relieve hot flashes in women based upon its ability to potentially modulate serotonin.

PURPOSE: This phase II trial is studying the side effects and how well s-adenosyl-L-methionine works in treating hot flashes in women with a history of breast cancer or those who do not wish to take estrogen due to a perceived increased risk of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the impact of SAMe on hot flash scores in women with a history of breast cancer or women who do not wish to take estrogen therapy for fear of increased risk of breast cancer.

II. To evaluate the toxicity of SAMe in this study population. III. To evaluate the effect of SAMe using quality-of-life (QOL) measures.

OUTLINE:

During the first week, participants will complete a daily, prospective hot flash diary and complete baseline questionnaires and will not be taking any study medication. After this baseline week, participants will receive oral s-adenosyl-L-methionine, 400 mg, once daily on days 8-14 and twice daily on days 15-49 in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of breast cancer (currently without malignant disease) or women who have no history of breast cancer but who wish to avoid estrogen due to a perceived increased risk of breast cancer
* Bothersome hot flashes (defined by their occurrence >= 14 times per week and of sufficient severity to make the patient desire therapeutic intervention)
* Presence of hot flashes for >= 1 month prior to registration
* Life expectancy >= 6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Ability to complete questionnaire(s) by themselves or with assistance
* Negative pregnancy test done =< 7 days prior to registration for women of childbearing potential only

Exclusion Criteria:

* Any of the following current (=< last 4 weeks) or planned therapies (tamoxifen, raloxifene, or aromatase inhibitors are allowed, but the patient must have been on a constant dose for >= 4 weeks and must not be expected to stop the medication during the study period): antineoplastic chemotherapy, androgens, estrogens, progestational agents, other herbal supplements, including soy, vitamin E, flaxseed, and megadose vitamins (herbal teas, multivitamins, and vitamin D are allowed), warfarin (1 mg of daily warfarin is allowed for central line patency), medications interacting with SAMe (antidepressants, monoamine oxidase (MAO) inhibitors, meperidine, dextromethorphan, pentazocine, tramadol, gabapentin, and levodopa)
* Pregnant women
* Nursing women
* Women of childbearing potential who are unwilling to employ adequate contraception
* Known allergy to SAMe
* Current use or use within the past 6 months of SAMe
* Clinically significant acute or chronic progressive or unstable neurologic, psychiatric, hepatic, renal, cardiovascular, respiratory, metabolic, or systemic disease precluding participation in the study
* History of bipolar disorder or Parkinsonism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five (45) subjects were recruited between October 2010 and January 2012 at Mayo Clinic.
Pre-assignment Details: Two subjects were ineligible and excluded from all analyses except adverse events summary.
Groups:
- SAMe: The first week of the study is a baseline week where data are being collected but study agent is not being taken. Patients then receive oral s-adenosyl-L-methionine, 400 mg, once daily on days 8-14 and twice daily on days 15-49 in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | SAMe
Started | 43
Completed | 34
Not Completed | 9
Not completed — Adverse Event | 4
Not completed — Refused Further Treatment | 5

BASELINE CHARACTERISTICS:
Arm/Group | SAMe
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 43
Tamoxifen Therapy [Number; unit: Participants]
  Yes | 8
  No | 35
Raloxifene Therapy [Number; unit: Participants]
  Yes | 0
  No | 43
Aromatase Inhibitor Therapy [Number; unit: Participants]
  Yes | 5
  No | 38
Average Hot Flashes per Day [Number; unit: Participants]
  2-3 | 3
  4-9 | 21
  >=10 | 19
Duration of Flash Symptoms (months) [Number; unit: Participants]
  <9 months | 5
  >=9 months | 38
Breast Cancer History [Number; unit: Participants]
  Yes | 18
  No | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Baseline in Average Hot Flash Activity (Score and Frequency)
Description: Hot flash score was defined as the number of mild hot flashes for the week plus two times the number of moderate hot flashes plus three times the number of severe hot flashes plus four times the number of very severe hot flashes. Hot flash frequency was defined as the average number of hot flashes per day for each week. Week 7 percent of baseline was calculated. The reduction in hot flash score and frequency can be calculated by subtracting the week 7 percent of baseline from 100 percent.
Time Frame: From baseline to week 7
Population: Analysis population includes only the subjects who have completed the quality of life self-assessment questionnaire.
Measure: Mean (95% Confidence Interval); unit: Percent of baseline
Arm/Group | SAMe
Number analyzed (Participants) | 31
Percent of baseline
  Week 7 percent of baseline for Hot Flash Score | 64.6 [49.2 to 80.0]
  Week 7 percent of baseline for Hot flash frequency | 67.4 [52.3 to 82.5]
Statistical Analysis 1: Comparison: SAMe; To determine whether any reduction in hot flash score is beyond what is expected with a placebo (20-25%). Reference: Sloan JA, et al. Methodologic lessons learned from hot flash studies. J Clin Oncol. Dec 1 2001;19(23):4280-4290; Test type: Superiority or Other; p = 0.0903, t-test, 1 sided — One sided t-test with 0.05 error rate was employed
Statistical Analysis 2: Comparison: SAMe; To determine whether any reduction in hot flash frequency is beyond what is expected with a placebo (20-25%). Reference: Sloan JA, et al. Methodologic lessons learned from hot flash studies. J Clin Oncol. Dec 1 2001;19(23):4280-4290; Test type: Superiority or Other; p = 0.1553, t-test, 1 sided — One sided t-test with 0.05 error rate was employed

2. Secondary Outcome: Change From Baseline to Week 7 for the Side Effect Questionnaire (SEQ)
Description: The side effect questionnaire (SEQ) consists of 15 items on a scale of 0 to 10 with 10 represents worse symptoms. Each item were reported as individual scores with all scores transposed to a 0-100 point percentage scale where 100 is the best quality of life (QOL) scores. Change from baseline to week 7 scores was calculated by subtracting the baseline scores from the scores at week 7. The positive change in scores indicates an improvement in QOL and negative change in scores indicates a decline in QOL.
Time Frame: Baseline and Week 7
Population: Includes all participants who initiated the study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAMe
Number analyzed (Participants) | 43
score on a scale
  Abnormal sweating: number analyzed (Participants) | 32
  Abnormal sweating | 25 (34.5)
  Trouble sleeping: number analyzed (Participants) | 32
  Trouble sleeping | 17.5 (30.7)
  Fatigue: number analyzed (Participants) | 29
  Fatigue | 11.7 (25.2)
  Muscle or joint aches/pain: number analyzed (Participants) | 32
  Muscle or joint aches/pain | 10 (20.6)
  Trouble concentrating: number analyzed (Participants) | 32
  Trouble concentrating | 7.5 (20.2)
  Swelling of hands/feet: number analyzed (Participants) | 32
  Swelling of hands/feet | 2.8 (18.9)
  Anxiousness: number analyzed (Participants) | 32
  Anxiousness | 2.8 (16.7)
  Constipation: number analyzed (Participants) | 32
  Constipation | 2.5 (25)
  Diarrhea: number analyzed (Participants) | 29
  Diarrhea | 1.4 (18.3)
  Headache: number analyzed (Participants) | 29
  Headache | 0 (16)
  Nausea: number analyzed (Participants) | 29
  Nausea | -1.4 (18.1)
  Lack of coordination: number analyzed (Participants) | 32
  Lack of coordination | -3.8 (14.8)
  Appetite: number analyzed (Participants) | 29
  Appetite | -4.1 (17.8)
  Dry mouth: number analyzed (Participants) | 29
  Dry mouth | -4.1 (22.4)
  Sleepiness: number analyzed (Participants) | 29
  Sleepiness | -15.5 (25.6)

3. Secondary Outcome: Change From Baseline to Week 7 for the Profile of Mood States (POMS)
Description: The Profile of Mood States (POMS) consists of 30 items on scale of 0 to 4 (0=not at all, 1=a little, 2=moderately, 3=quite a bit and 4=extremely). The POMS was scored according to its specific scoring algorithm resulting in a total score and six subscale scores (anger/hostility, confusion/bewilderment, depression/dejection, fatigue/inertia, tension/anxiety, and vigor/activity). All scores were transposed to a 0-100 point percentage scale where 100 is the best quality of life (QOL) scores. Change from baseline to week 7 scores was calculated by subtracting the baseline scores from the scores at week 7. The positive change in scores indicates an improvement in QOL and negative change in scores indicates a decline in QOL.
Time Frame: Baseline and Week 7
Population: Includes all participants who initiated the study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAMe
Number analyzed (Participants) | 43
score on a scale
  POMS total: number analyzed (Participants) | 30
  POMS total | 3.0 (7.8)
  Fatigue/inertia: number analyzed (Participants) | 30
  Fatigue/inertia | 10.9 (18.7)
  Anger/hostility: number analyzed (Participants) | 30
  Anger/hostility | 2.8 (10.1)
  Tension/anxiety: number analyzed (Participants) | 30
  Tension/anxiety | 2.3 (10.8)
  Confusion/bewilderment: number analyzed (Participants) | 30
  Confusion/bewilderment | 1.2 (10.6)
  Depression/dejection: number analyzed (Participants) | 30
  Depression/dejection | 0.7 (8.8)
  Vigor/activity: number analyzed (Participants) | 30
  Vigor/activity | 0.5 (13.9)

4. Secondary Outcome: Change From Baseline to Week 7 for the Hot Flash Related Daily Interference Scale (HFRDIS)
Description: The Hot Flash Related Daily Interference Scale (HFRDIS) consists of 10 items on scale of 0 to 10 with 0 represents do not interfere and 10 represents completely interferes. An average of the scores of the 10 individual items was calculated for the HFRDIS total score. Each individual item were reported as individual scores. All scores were transposed to a 0-100 point percentage scale where 100 is the best quality of life (QOL) scores. Change from baseline to week 7 scores was calculated by subtracting the baseline scores from the scores at week 7. The positive change in scores indicates an improvement in QOL and negative change in scores indicates a decline in QOL.
Time Frame: Baseline and Week 7
Population: Includes all participants who initiated the study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAMe
Number analyzed (Participants) | 43
score on a scale
  HFRDIS total: number analyzed (Participants) | 31
  HFRDIS total | 8.6 (14.4)
  Mood: number analyzed (Participants) | 31
  Mood | 13.9 (16.3)
  Sleep: number analyzed (Participants) | 32
  Sleep | 21.6 (30.0)
  Concentration: number analyzed (Participants) | 32
  Concentration | 12.8 (21.3)
  Overall QOL: number analyzed (Participants) | 32
  Overall QOL | 7.8 (21.1)
  Enjoyment of life: number analyzed (Participants) | 32
  Enjoyment of life | 5.9 (17.4)
  Social activities: number analyzed (Participants) | 32
  Social activities | 5.3 (17.0)
  Leisure activities: number analyzed (Participants) | 32
  Leisure activities | 4.7 (15.2)
  Work: number analyzed (Participants) | 32
  Work | 4.4 (19.3)
  Relationships with others: number analyzed (Participants) | 32
  Relationships with others | 3.4 (15.6)
  Sexuality: number analyzed (Participants) | 32
  Sexuality | 2.8 (23.7)

5. Secondary Outcome: Number of Patients Who Reported Grade 3 Adverse Events
Description: Adverse events were assessed per NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: Week 1 to Week 7
Population: All participants who enrolled to the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | SAMe
Number analyzed (Participants) | 45
Participants
  Insomnia | 2
  Neoplasms: benign, malignant, unspecified | 1

ADVERSE EVENTS:
Description: All participants who enrolled to the trial.
Arm/Group | SAMe
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 41/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAMe (N=45)
Insomnia (Psychiatric disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAMe (N=45)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Bloating (Gastrointestinal disorders) | 23 (76)
Diarrhea (Gastrointestinal disorders) | 11 (26)
Nausea (Gastrointestinal disorders) | 16 (28)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Allergic reaction (Immune system disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 36 (143)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes